CLINICAL TRIAL: NCT04346355
Title: An Open-label Randomized Multicenter Study to Evaluate the Efficacy of Early Administration of Tocilizumab (TCZ) in Patients With COVID-19 Pneumonia
Brief Title: Efficacy of Early Administration of Tocilizumab in COVID-19 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on interim analysis for futility and given an enrolment rate almost nil
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-TCZ-COVID-19; 2020-001386-37 (EudraCT Number)
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — tocilizumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Tocilizumab within 8 hours from entering the study + standard of care; 8 mg/kg IV up to a maximum of 800 mg with repetition of the same dosage after 12 hours
  Interventions: Drug: Tocilizumab
- Control Arm (Other): Standard of care; In the event of aggravation of COVID-19 pneumonia, according to protocol criteria, participants will receive 8 mg/kg IV up to a maximum of 800 mg with repetition of the same dosage after 12 hours
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — In case of aggravation of COVID-19 pneumonia, according to protocol criteria, participants will receive 8 mg/kg IV up to a maximum of 800 mg with repetition of the same dosage after 12 hours
  Other Names: Standard of care

SUMMARY:
The clinical study aims at assessing whether early administration of Tocilizumab compared to late administration of Tocilizumab can reduce the number of patients with COVID-19 pneumonia who require mechanical ventilation. The clinical study includes patients with recent-onset COVID-19 pneumonia who require hospital care, but not invasive or semi-invasive mechanical ventilation procedures.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Informed consent for participation in the study
* Real time polymerase chain reaction (PCR) diagnosis of Sars-CoV2 infection
* Hospitalization due to clinical / instrumental diagnosis (high resolution chest CT scan or chest x-ray or pulmonary ultrasound)
* Presence of acute respiratory distress syndrome with arterial partial pressure of oxygen / fraction of inspired oxygen (PaO2 / FiO2) between 200 and 300 mm/Hg
* Presence of exaggerated inflammatory response defined by the presence of at least 1 of the following criteria:
* At least one body temperature measurement >38° C in the past two days;
* Serum CRP greater than or equal to 10 mg/dl;
* CRP increase of at least twice the basal value

Exclusion Criteria:

* Patients with respiratory distress syndrome with arterial partial pressure of oxygen / fraction of inspired oxygen (PaO2 / FiO2) <200 mm/Hg or
* Patients in non-invasive ventilation or
* Patients in invasive ventilation or presence of shock or presence of concomitant organ failure that requires admission to the Intensive Care Unit
* Severe heart and kidney failure
* Pregnant or breastfeeding patient
* Patient who, in the opinion of the clinician or by the patient's express will, will not go to intensive care regardless of the evolution of the lung picture.
* Known hypersensitivity to TCZ or its excipients
* Patient being treated with immuno-depressors or anti-rejection drugs
* Known active infections or other clinical conditions that contraindicate TCZ and cannot be treated or resolved according to the physician's judgment
* glutamate-pyruvate transaminase (GPT) or glutamine oxaloacetic transaminase (GOT) > 5 times the upper limit of the norm
* Neutrophils <500 /mmc
* Platelets <50.000 /mmc
* Diverticulitis or intestinal perforation
* Suspicion of latent tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Entry into Intensive Care with invasive mechanical ventilation or death from any cause or clinical aggravation | two weeks from participants' allocation to study arm
  Entry into Intensive Care with invasive mechanical ventilation or death from any cause or clinical aggravation documented by the finding of a PaO2 / FiO2 ratio <150mm / Hg confirmed by a second arterial blood gas (ABG) measurement within four hours

SECONDARY OUTCOMES:
Death from any cause | Two weeks from participants' allocation to study arm
  Death
Tocilizumab toxicity | Two weeks from participants' allocation to study arm
  Adverse events (AE) classified according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale
Levels of interleukin-6 and C-reactive protein (CRP) and their correlation with the effectiveness of the treatment | Two weeks from participants' allocation to study arm
  Levels of ferritin, lactate dehydrogenase and D-dimer and their correlation with the effectiveness of the treatment
Evaluate the progress of the PaO2 / FiO2 ratio | Two weeks from participants' allocation to study arm
  Changes from baseline of the PaO2 / FiO2 ratio
Evaluate the trend over time of the lymphocyte count | Two weeks from participants' allocation to study arm
  Changes from baseline of the lymphocyte count

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Salvarani, M.D., Study Director — Azienda Unità Sanitaria Locale-IRCCS di Reggio Emilia; Massimo Costantini, Ph.D., Study Director — Azienda Unità Sanitaria Locale-IRCCS di Reggio Emilia
Locations (25):
- Italy (25):
  - Ospedale di Guastalla, Guastalla, RE
  - Azienda Unità Sanitaria Locale-IRCCS di Reggio Emilia, Reggio Emilia, RE
  - Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Policlinico Sant'Orsola Malpighi, Bologna
  - ASST Cremona, Cremona
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Azienda Ospedaliero Universitaria Ferrara, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Evangelico Internazionale di Genova, Genova
  - Azienda Sociosanitaria ASL 1 ,Imperia, Imperia
  - Azienda Sociosanitaria ASL 5 La Spezia, La Spezia
  - ASST Mantova - Ospedale Carlo Poma, Mantova
  - IRCCS Istituto Auxologico Italiano Milano, Milan
  - Azienda Ospedaliero-Universitaria "Maggiore della Carità" di Novara, Novara
  - Ospedali Riuniti Padova Sud - ULSS 6 Euganea, Padua
  - Azienda Ospedaliero-Universitaria Parma, Parma
  - Azienda Unità Sanitaria Locale di Piacenza, Piacenza
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - AO Ordine Mauriziano di Torino, Torino
  - ASST Bergamo Ovest -Treviglio, Treviglio
  - AULSS 2 Marca Trevigiana, Treviso
  - AULSS2 Marca Trevigiana - Ospedale Vittorio Veneto, Treviso
  - AULSS 3 Serenissima Ospedale "Dell'Angelo", Venezia
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
  - IRCCS Sacro Cuore Don Calabria, Verona

REFERENCES:
- [Derived] Salvarani C, Dolci G, Massari M, Merlo DF, Cavuto S, Savoldi L, Bruzzi P, Boni F, Braglia L, Turra C, Ballerini PF, Sciascia R, Zammarchi L, Para O, Scotton PG, Inojosa WO, Ravagnani V, Salerno ND, Sainaghi PP, Brignone A, Codeluppi M, Teopompi E, Milesi M, Bertomoro P, Claudio N, Salio M, Falcone M, Cenderello G, Donghi L, Del Bono V, Colombelli PL, Angheben A, Passaro A, Secondo G, Pascale R, Piazza I, Facciolongo N, Costantini M; RCT-TCZ-COVID-19 Study Group. Effect of Tocilizumab vs Standard Care on Clinical Worsening in Patients Hospitalized With COVID-19 Pneumonia: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jan 1;181(1):24-31. doi: 10.1001/jamainternmed.2020.6615. PMID 33080005